CLINICAL TRIAL: NCT06418932
Title: Compression Therapy of the Lower Limbs in Patients With Decompensated Heart Failure and Predominant Systemic Tissue Congestion
Brief Title: Compression Therapy of the Lower Limbs in Patients With Decompensated Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMPRESSION-HF
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to standard treatment (parenteral administration of furosemide) versus parenteral administration of furosemide plus lower limb compression therapy for a maximum of 72 hours. The dose of furosemide in all participants will be based on the clinical judgment of the responsible health professional.
Who Masked: Participant, Investigator
Masking Description: Sham procedure. Blinded to treatment allocation. The investigator and the patients will be blinded to treatment assignments. For this purpose, a restraint system will be used which will be applied to the lower limbs and will mask the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive (Experimental): Compressive therapy of the lower limbs plus parenteral administration of diuretics
  Interventions: Device: UrgoK2 / UrgoK2 Lite
- Control (Active Comparator): Parenteral diuretics alone
  Interventions: Other: Controll

INTERVENTIONS:
Device: UrgoK2 / UrgoK2 Lite — Multicomponent compressive bandage system consisting of an internal bandage of short traction and an external cohesive bandage of long traction, with pressure indicators on both bandages, which provides a sustained ankle pressure of ~20/40mmHg.
  Arms: Compressive
Other: Controll — Administration of parenteral diuretics only
  Arms: Control

SUMMARY:
Randomized 1:1 multicenter double-blind clinical investigation evaluating the efficacy and safety of compression therapy of the lower limbs plus parenteral administration of diuretics vs. administration of parenteral diuretics alone (standard treatment) in patients with decompensated HF and predominantly systemic tissue congestion and absence of intravascular systemic congestion.

Patients will be assigned to standard treatment (parenteral administration of furosemide) versus parenteral administration of furosemide plus lower limb compression therapy for up to 72 hours. The dose of furosemide in all participants will be based on the clinical judgment of the responsible healthcare professional.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patient with clinical judgment of acute decompensated heart failure in the first 96 hours from the start of parenteral diuretic treatment.
* Patient treated with furosemide at least 40 mg in the last 24 hours.
* NT-proBNP levels>1000 pg/ml at least 1 time since the onset of decompensation.
* Presence of tibio-malleolar edema at least grade II/IV at the time of inclusion.
* Inferior vena cava (IVC) diameter on ultrasonography ≤21 mm at the time of the "screening" visit.

Exclusion Criteria:

* Being admitted to the Intensive Care Unit.
* Renal transplant, chronic renal failure stage 5 (eGFR <15 ml/min/1.73m2) or being included in dialysis program (peritoneal/hemodialysis) or in need of ultrafiltration.
* Absence of peripheral pulses.
* Ankle brachial index (ABI) <0.9.
* History of severe peripheral artery disease.
* Previous intolerance to compressive bandaging.
* HF secondary to acute myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Natriuresis | 24 hours
  Changes in natriuresis at 24 hours after randomization.
Weight | 24 hours
  Changes in weight at 24 hours after randomization

SECONDARY OUTCOMES:
Diameter of the lower limbs | 72 hours
  Changes in the diameter of the lower limbs (at 5 and 10 cm from the ankles) at 24 and 72 hours after randomization.
Congestion score | 72 hours
  Changes in clinical congestion score at 24 and 72 hours
Inferior vena cava diameter | 72 hours
  Changes in inferior vena cava diameter at 3, 24 and 72 hours
NT-proBNP | 72 hours
  Changes in circulating levels of the N-terminal portion of B-type natriuretic pro-peptide (NT-proBNP) at 72 hours.
CA125 | 15±3 days
  Changes in circulating levels of carbohydrate antigen 125 (CA125) at 15±3 days
Doses of furosemide | 72 hours
  Doses of furosemide equivalents used in the first 72 hours after randomization
Time to oral administration. | 72 hours
  Time to switch from diuretics to oral administration

OTHER OUTCOMES:
Tolerance | 72 hours
  Percentage of patients in whom tolerance of the compressive bandage is achieved at 24 and 72 hours
eGFR | 72 hours
  Estimated glomerular filtration rate (eGFR) at 72 hours
Electrolyte disturbances | 72 hours
  Electrolyte disturbances at 72 hours (hyponatremia: <135 mmo/l, hypernatremia>150 mmo/l, hypokalemia<3.5 mmo/l and hyperkalemia>5 mmo/l)
Clinical adverse events | 30 days
  Clinical adverse events at 30 days total and cardiovascular, with special emphasis on cardiovascular death and HF decompensation

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital de Denia, Denia, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital General de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No